CLINICAL TRIAL: NCT06034847
Title: Treatment of Persistent Distal Occlusion After Successful Proximal Recanalization in Thrombectomy
Acronym: 2BE3
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-11741
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Stroke, Acute Thrombotic
Keywords: Large vessel occlusion; Persistent distal occlusion; Mechanical thrombectomy; Intra-arterial thrombolytics
MeSH Terms: conditions — Thrombotic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conservative management (Active Comparator): Mechanical thrombectomy of large vessel occlusions with or without administration of IV thrombolytics
  Interventions: Device: Mechanical thrombectomy in proximal large vessels
- Rescue therapy (Active Comparator): In addition to conservative management, rescue therapy in distal occlusions consisting of either mechanical thrombectomy with small stent retrievers with or without contact aspiration, or intra-arterial pharmacotherapy with tPA (tissue Plasminogen Activator), uPA (urokinase Plasminogen Activator) or tenecteplase.
  Interventions: Device: Mechanical thrombectomy in proximal large vessels; Device: Rescue mechanical thrombectomy in distal vessels

INTERVENTIONS:
Device: Mechanical thrombectomy in proximal large vessels — mechanical thrombectomy with retrievable stents to remove clots in proximal large vessels, combined or not with distal aspiration, combined or not with IV thrombolytics
Device: Rescue mechanical thrombectomy in distal vessels — In addition to mechanical thrombectomy in proximal large vessels, mechanical thrombectomy in distal vessels with small stent retrievers combined or not with contact aspiration, or intra-arterial perfusion of thrombolytics such as tPA or uPA or tenecpeplase
  Arms: Rescue therapy

SUMMARY:
In stroke patients, mechanical thrombectomy is now the standard of care when the stroke is due to large proximal cerebral vessel occlusion. The purpose of the 2BE3 trial is to test whether adjunct rescue treatment of persisting distal occlusions after successful proximal recanalization of the large vessel occlusion can be proposed as an additional intervention to restore reperfusion of affected stroke tissue and improve clinical outcomes.

The rescue therapies will be either mechanical (small stent retrievers and/or small aspiration catheters) or pharmacological (infusion of intra-arterial thrombolytics).

Patients will be randomized to conservative management (mechanical thrombectomy with or without IV thrombolytics of large proximal vessels) or rescue therapy (mechanical or pharmacological interventions in distal vessels in addition to conservative management). Each patient will be followed for 3 months post-intervention.

The data collected will be clinical assessments and angiographic imaging to evaluate the reperfusion state.

DETAILED DESCRIPTION:
The purpose of the 2BE3 trial is to provide a clinical trial context for the use of rescue therapy (mechanical or pharmacological therapies) in patients with persistent distal occlusions after treatment of large vessel occlusions with mechanical thrombectomy and IV thrombolytics. The main hypothesis is that rescue therapy with mechanical or pharmacological therapies, compared with conservative management would result in improved clinical and reperfusion scores at 90 days.

The extent of reperfusion is an interesting therapeutic target because reperfusion status is a strong indicator of clinical outcome: grades of better reperfusion are incrementally associated with better clinical outcomes. Despite increased expertise of neuro-interventional teams and the evolution in thrombectomy devices, incomplete reperfusion occurs in almost half of patients undergoing treatment of large vessel occlusions. Thus, complementary treatments targeting distal occlusions and known as "rescue therapy" have been introduced to reach complete or near complete reperfusion.

The devices and techniques proposed as rescue therapies include small stent retrievers, small aspiration catheters and intra-arterial thrombolytics. Case studies and registries have shown high reperfusion rates and low rates of periprocedural complications; however, there is lack of randomized data to show the impact of rescue therapies on patient outcomes and safety compared to conservative management (treatment of large vessel occlusions only). A randomized clinical trial is therefore needed.

The 2BE3 trial is a simple randomized trial designed to be integrated into daily clinical practice. It will address whether rescue therapies truly offer a safe and more effective alternative to conservative management. Selection criteria are loose in order to be of use to most patients. Endpoints are simple, clinical, meaningful, valuable and resistant to bias. It includes no extra risk or cost of visits beyond what is required in routine care.

The design is multicenter, prospective, randomized, controlled, open-label study with blinded evaluation (PROBE design). The study population is acute ischemic stroke patients with persistent distal occlusions after treatment of large vessel occlusion with mechanical thrombectomy and/or intravenous thrombolysis. The total number of patients will be 300, 150 in each arm, each followed for 3 months post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* any patient with a large vessel occlusion in the M1 or M2 segment of the MCA (Middle Cerebral Artery), supraclinoid ICA (Internal Carotid Artery), or basilar artery who is a candidate for thrombectomy
* with a persistent distal occlusion in M2-M4, A1-A5, P1-P5 after successful recanalization of the proximal clot with mechanical thrombectomy and/or IV thrombolysis

Exclusion Criteria:

* poor 3 month prognosis from comorbidities
* evidence of active bleeding on examination
* recent surgery with a significant risk of bleeding
* VKA (Vitamin K Antagonists) oral anticoagulation with INR (International Normalized Ratio) - > 1.7
* curative heparin or direct oral anticoagulants in previous 48 hours
* platelet count < 100 000/mm3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Rate of modified Rankin Scale score of 0-2. The modified Rankin score goes from 0 (no symptoms) to 6 (death). Higher scores mean a worse outcome | 90 days
  proportion of patients with a modified Rankin Scale score of 0-2

SECONDARY OUTCOMES:
score on the modified Rankin Scale. The modified Rankin score goes from 0 (no symptoms) to 6 (death). Higher scores mean a worse outcome | 90 days
  score on the modified Rankin Scale
Rate of functional independence | 90 days
  Functional independence is defined as a modified Rankin Scale score of 0-2
Change in NIHSS (National Institutes of Health Stroke Score) score. The scale goes from 0 to 42; higher scores indicated worse outcomes. | 24 hours
  Difference between the NIHSS score at Registration and at 24 hours post-intervention
Rate of NIHSS (National Institutes of Health Stroke Score) score improvement. The scale goes from 0 to 42; higher scores indicated worse outcomes. | 24 hours
  Rate of decrease of 4 points or more in NIHSS score
Rate of improved global ipsilateral hemispheric reperfusion | at end of procedure
  blinded assessment of reperfusion on angiogram as measured by the modified TICI (Thrombolysis in Cerebral Infarction) scale. The scale goes from 0 to 3; higher scores indicate better outcomes
Rate of reperfusion | at end of procedure
  assessed by the modified TICI (Thrombolysis in Cerebral Infarction) scale on angiogram. The scale goes from 0 to 3; higher scores indicate better outcomes
Rate of complete reperfusion | at end of procedure
  a modified TICI (Thrombolysis in Cerebral Infarction) score of 3 on angiogram. The scale goes from 0 to 3; higher scores indicate better outcomes
Procedure time | at end of procedure
  elapsed time from arterial puncture to last angiogram
Number of thrombectomy passes | at end of procedure
  Number of thrombectomy passes to achieve final reperfusion
Mortality rate | 24 hours and 90 days
  Rate of mortality
Rate of procedural complications | at end of procedure
  defined as: vascular perforation, arterial dissection, new territory emboli, access site complication requiring surgical repair, subarachnoid hemorrhage
Rate of symptomatic intracerebral hemorrhage | 24 hours
  hemorrhage on CT or MRI according to the Heidelberg classification associated with a 4 point or greater worsening on the NIHSS score. The Heidelberg classification goes from 1 to 3d; higher scores indicate worse outcomes.
Rate of any intracranial hemorrhage | 24 hours
  hemorrhage on CT or MRI according to the Heidelberg classification. The Heidelberg classification goes from 1 to 3d; higher scores indicate worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Iancu, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- CHUM - Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
there is no plan to share individual participant data